CLINICAL TRIAL: NCT03863054
Title: An Observational Clinical Trial Examining the Effect of Topical Oxygen Therapy (NATROX™) on the Rates of Healing of Chronic Diabetic Foot Ulcers
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/2355
Record Dates: First submitted 2019-03-04; First posted 2019-03-05 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Foot Ulcer; Non-healing Wound
Keywords: Topical Oxygen; Wound Management
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- >40% wound area reduction after 1 month: Subjects to continue with standard practice for the next 12 weeks, or until the wound has completely healed.
- <40% wound area reduction after 1 month: Subjects to be fitted with NATROX™ after 1 month, over a period of 12 weeks or until the wound has completely healed.
  Interventions: Device: NATROX™ Topical Oxygen Therapy System

INTERVENTIONS:
Device: NATROX™ Topical Oxygen Therapy System — A small battery-powered electrochemical "oxygen generator" to concentrate atmospheric oxygen and feed to wound site through a dressing-like "oxygen distribution system"
  Groups: <40% wound area reduction after 1 month

SUMMARY:
This study aims to evaluate the effectiveness of NATROX™ Topical Oxygen Wound Therapy for subjects with non-healing foot ulceration. Subjects will be treated with standard care for 4 weeks. If the wound is not reduced by more than 40%, NATROX™ will be applied for the next 12 weeks. Throughout the study period, wound measurements will be taken to measure wound reduction.

DETAILED DESCRIPTION:
Diabetes and its attendant complications are increasing year on year. A number of macro- and micro-circulatory changes occur as a result of long standing or poorly controlled diabetes. These, often in association with either loss of lower limb sensation, or mechanical changes in the foot architecture, can lead to the formation of foot ulcers. These can be hard to heal because of the changes in the diabetic foot described above, as well as an increased incidence of infection in this population. Invasive or ascending infection through these breaks in the skin can lead to tissue loss, which may range from a single toe to major amputation below or above the knee. Major limb amputation has a profound effect on patient's quality of life, as well as a significant economic impact on the health and social care budget. Caring for diabetic foot ulcers, and the complications of this, have a cost of around S$1.2 billion per annum, which has become a focus of public health concern in Singapore recently.

The concept of increasing the oxygen concentration in healing wounds developed originally with hyperbaric oxygen therapy, and from the fact that oxygen is one of the most essential elements used during cellular metabolism. Poor tissue oxygenation, as is often seen in diabetic foot ulcers, is a significant impediment to cellular activity, and is therefore very likely to impair wound healing.

The NATROX™ topical oxygen therapy system developed by Inotec AMD Limited employs a small battery-powered electrochemical "oxygen generator" to concentrate atmospheric oxygen and feed the pure, moist, oxygen at a rate of around 13ml/hour through a fine, soft, tube to a dressing-like "oxygen distribution system" that is placed over the wound and is held in place by a conventional dressing. The oxygen generator is worn in a holster on the waist or above the calf, or is placed in a trouser pocket, thus enabling the patient to enjoy normal mobility (hence "ambulatory") while receiving continuous treatment.

The very significant costs of treatment of diabetic foot ulcers and the impact of amputations on quality of life and life expectancy, suggest that Natrox™ treatment is likely to be cost effective, a conclusion that was evident from the brief independent health economics study linked to the project. To date, no Asian study looking at whether the device is efficacious in a multi-racial population like Singapore. The vessels in Asians are generally smaller and the micro circulation is generally more diseased than our Caucasian counterparts because of the higher incidence of diabetes. This technology could be ideal for such patients and improve our limb salvage rates. After revascularization and control of infection, there is little alternative if the wound does not heal apart from further wound debridement or major amputation. This study may show us which Diabetic Foot Ulcers or wounds are likely to respond to topical oxygen and what effect it has on the patient per se in terms of pain relief and improvement of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* A diabetic foot ulcer greater than 12 weeks and less than 18 months in duration
* Minor amputation sites <50% healed in 4 weeks (the use of negative pressure wound therapy to optimize the wound bed is allowable)
* 4 weeks of standard of care at the hospital based diabetic foot clinic or in a specialist community diabetic podiatry clinic prior to entry into the open registry
* No planned revascularization (endovascular or open surgery) within 4 weeks following revascularization being performed)
* Ongoing active chemical or sharp wound debridement prior to and during the application of NATROX™
* No limit on level of ischemia, either high or low. The extent of arterial disease will be documented by angiogram or duplex ultrasound and toe blood pressure
* The subject is 21 years of age or older
* The subject is willing to complete >75% of follow-up evaluations required by the study protocol
* The subject is able to abstain from any other clinical trial for the duration of the study
* The study is able to read and understand instructions and give voluntary written informed consent
* The subject is able and willing to follow the protocol requirements

Exclusion Criteria:

* Inability to comply with the dressing regime or manage the NATROX™ device
* Disseminated malignancy
* Subjects with a >1 year life expectancy
* Subjects with an ulcer which is <0.5cm2 or >50cm2
* Subjects who is dialysis dependent for less than 1 year (i.e. subject is eligible for study if has CKD/ESRF and is on dialysis for >1year)
* The subject has an invasive soft tissue infection at the time of baseline assessment, requiring oral or intravenous antibiotic therapy.
* Exposed bone without soft tissue or granulation tissue across the surface
* Acute osteomyelitis (stable, chronic osteomyelitis is allowable, including those maintained on oral antibiotics, as long as there is no planned intervention)
* Pregnant/lactating females (self-reported or tested, as per institutional requirements)
* Glycated haemoglobin HbA1C of >12mmol mol-1
* Subject who have evidence of connective tissue disorders (e.g. vasculitis or rheumatoid arthritis) under active treatment
* The subject is unable to follow the protocol
* The subject has other concurrent conditions that in the opinion of the investigator may compromise subject safety
* The patient is a vulnerable or protected adult
* The patient is unable to provide informed consent
* Diabetic foot ulcer is connected to a sinus wound

Ages: 21 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with non-healing Diabetic Foot Ulcers that has been persistent for more than 3 months, or less than 50% healing observed within 1 month for amputation sites.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage change in ulcer size | 12 weeks after NATROX™ fitted
  after 12 weeks of NATROX™ therapy, relative to baseline measurement

SECONDARY OUTCOMES:
Absolute Closure Number | 16 weeks after last patient enrolled
  Total number of patients with wounds that completely healed at the end of study period
Wound Closure Rate relative to the 4-week run in period | 16 weeks after last patient enrolled
  Number of wounds 100% healed at the end of 4 week run-in
Number of dressing episodes during the study period | 16 weeks after enrolment
Number of infection episodes | 16 weeks after enrolment
Diabetic Foot Ulcer Scale | Baseline (week 0), Week 4, Week 8, Week 12 and Week 16 post enrolment
  To assess quality of life
Pain at wound site | Baseline (week 0), Week 4, Week 8, Week 12 and Week 16 post enrolment
  Assessed using a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Tang Tjun Yip, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blackman E, Moore C, Hyatt J, Railton R, Frye C. Topical wound oxygen therapy in the treatment of severe diabetic foot ulcers: a prospective controlled study. Ostomy Wound Manage. 2010 Jun;56(6):24-31. PMID 20567051
- [Background] Driver VR, Yao M, Kantarci A, Gu G, Park N, Hasturk H. A prospective, randomized clinical study evaluating the effect of transdermal continuous oxygen therapy on biological processes and foot ulcer healing in persons with diabetes mellitus. Ostomy Wound Manage. 2013 Nov;59(11):19-26. PMID 24201169
- [Background] Gordillo GM, Sen CK. Evidence-based recommendations for the use of topical oxygen therapy in the treatment of lower extremity wounds. Int J Low Extrem Wounds. 2009 Jun;8(2):105-11. doi: 10.1177/1534734609335149. PMID 19443899
- [Background] Hirsh F, Berlin SJ, Holtz A. Transdermal oxygen delivery to diabetic wounds: a report of 6 cases. Adv Skin Wound Care. 2009 Jan;22(1):20-4. doi: 10.1097/01.ASW.0000343722.22943.40. PMID 19096280
- [Background] Gordillo GM, Roy S, Khanna S, Schlanger R, Khandelwal S, Phillips G, Sen CK. Topical oxygen therapy induces vascular endothelial growth factor expression and improves closure of clinically presented chronic wounds. Clin Exp Pharmacol Physiol. 2008 Aug;35(8):957-64. doi: 10.1111/j.1440-1681.2008.04934.x. Epub 2008 Apr 21. PMID 18430064
- [Background] Driver VR, Reyzelman A, Kawalec J, French M. A Prospective, Randomized, Blinded, Controlled Trial Comparing Transdermal Continuous Oxygen Delivery to Moist Wound Therapy for the Treatment of Diabetic Foot Ulcers. Ostomy Wound Manage. 2017 Apr;63(4):12-28. PMID 28448266
- [Background] Tawfick WA, Sultan S. Technical and clinical outcome of topical wound oxygen in comparison to conventional compression dressings in the management of refractory nonhealing venous ulcers. Vasc Endovascular Surg. 2013 Jan;47(1):30-7. doi: 10.1177/1538574412467684. Epub 2012 Dec 5. PMID 23223182
- [Background] Niederauer MQ, Michalek JE, Armstrong DG. A Prospective, Randomized, Double-Blind Multicenter Study Comparing Continuous Diffusion of Oxygen Therapy to Sham Therapy in the Treatment of Diabetic Foot Ulcers. J Diabetes Sci Technol. 2017 Sep;11(5):883-891. doi: 10.1177/1932296817695574. Epub 2017 Feb 15. PMID 28654304
- [Background] Tawfick W, Sultan S. Does topical wound oxygen (TWO2) offer an improved outcome over conventional compression dressings (CCD) in the management of refractory venous ulcers (RVU)? A parallel observational comparative study. Eur J Vasc Endovasc Surg. 2009 Jul;38(1):125-32. doi: 10.1016/j.ejvs.2009.03.027. Epub 2009 May 22. PMID 19464933
- [Background] Woo KY, Coutts PM, Sibbald RG. Continuous topical oxygen for the treatment of chronic wounds: a pilot study. Adv Skin Wound Care. 2012 Dec;25(12):543-7. doi: 10.1097/01.ASW.0000423439.62789.90. PMID 23151764
- [Background] Yu J, Lu S, McLaren AM, Perry JA, Cross KM. Topical oxygen therapy results in complete wound healing in diabetic foot ulcers. Wound Repair Regen. 2016 Nov;24(6):1066-1072. doi: 10.1111/wrr.12490. Epub 2016 Nov 2. PMID 27733020
- [Background] Hayes PD, Alzuhir N, Curran G, Loftus IM. Topical oxygen therapy promotes the healing of chronic diabetic foot ulcers: a pilot study. J Wound Care. 2017 Nov 2;26(11):652-660. doi: 10.12968/jowc.2017.26.11.652. PMID 29131746
- [Background] Mani R. Topical oxygen therapy for chronic wounds: a report on the potential of NATROX™ - a new device for delivering enriched oxygen to chronic wounds. Journal of Wound Technology 9:28-30, 2010
- [Derived] Tang TY, Mak MYQ, Yap CJQ, Boey JEC, Chan SL, Soon SXY, Ishak IAB, Lee RWL, Soh XJ, Goh WX. An Observational Clinical Trial Examining the Effect of Topical Oxygen Therapy (Natrox) on the Rates of Healing of Chronic DiAbetic Foot Ulcers (OTONAL Trial). Int J Low Extrem Wounds. 2024 Jun;23(2):326-337. doi: 10.1177/15347346211053694. Epub 2021 Nov 6. PMID 34747267